Title: Heel Wedges and Carbon Fiber Custom Dynamic Orthoses to Control Knee Biomechanics

NCT Number: NCT05209360

**Date:** October 19, 2023

#### **Study Protocol**

#### Purpose and Procedures:

The primary purpose of this line of research is to investigate the effects of combined carbon fiber custom dynamic orthosis (CDO) and medial-lateral wedge use on biomechanics during gait in an effort to reduce unilateral knee compartment loading. In this research study, pilot data will be collected from a cohort of healthy adult participants with no history of lower limb injuries or functional deficits. Participants will be evaluated using a series of study measures under each of the four conditions; without a brace (NoCDO), with a brace and no wedge (CDO), with a brace and a medial wedge placed in the shoe (Medial), and with a brace and a lateral wedge placed in the shoe (Lateral). Testing order will be randomized for each participant. Participants will walk on a level-ground walkway at self-selected and controlled speeds. Physical performance measures will incorporate tests of agility, speed, and lower limb power to ensure that the device and wedge don't negatively affect physical function. Questionnaires will be used to evaluate participants' pain and perception of comfort and smoothness for each condition.

#### Objectives and Specific Aims:

Specific Aim 1: Determine the effect of CDO alignment on lower limb mechanics during gait in a cohort of healthy individuals.

Specific Aim 2: Determine the effect of CDO alignment on physical function and patient reported outcomes in a cohort of healthy individuals.

#### Background and Significance:

Osteoarthritis (OA) affects nearly 27 million people in the United States alone, and accounts for approximately \$2,600 - \$7,500 in out of packet expenses each year.[2] Knee OA can affect the medial, the lateral, or both compartments of knee. Treatment of OA can include a number of options such as medial-lateral wedging under the foot, knee orthoses, or ankle foot orthoses (AFOs). In the case of unilateral medial compartment knee OA unloader knee braces are commonly used to decrease knee adduction moments in an attempt to offload the knee. Similar efforts have been completed with the use of medial-lateral wedge placed in the shoe under the heel of the foot. Wedging was shown to stabilize biomechanics over time, preventing increases in knee adduction moment over a one-year period compared to neutral wedging. In another study, an ankle foot orthosis with a lateral strut was used in an effort to move the center of pressure position, thereby altering frontal plane knee moment. Use of this AFO resulted in improved pain, stiffness, and physical function scores when assed using the Western Ontario and McMasters Universities Arthritics Index (WOMAC).

CDOs consist of a cuff that falls just below the knee, a carbon fiber spring that runs the length of the calf and bends to store and return energy during gait, and a footplate the acts as a lever arm to bend the posterior strut. CDOs stabilize the ankle, and this may allow for greater affects at the knee when frontal plane alignment is adjusted. Similar to application of medial-lateral heel wedges in the shoe, placing medial-lateral wedges under a CDO may also reduce knee adduction moments. The purpose of this study is to determine if medial-lateral wedging combined with CDO use alters knee biomechanics, physical function, and patient reported outcomes.

## Inclusion Exclusion Criteria:

## Patient Inclusion Criteria

- 1) Between the ages of 18 and 45
- 2) Healthy without current complaint of lower extremity pain, spine pain, open wounds or active infections, or medical or neuromusculoskeletal disorders that have limited their participation in work or exercise in the last 6 months
- 3) Able to hop without pain

- 4) Able to perform a full squat without pain
- 5) Ability to speak and understand English

## Patient Exclusion Criteria

- 1) Medical or neuromusculoskeletal disorders that have limited their participation in work or exercise in the last 6 months
- 2) Diagnosed with a moderate or severe brain injury
- 3) Lower extremity injury resulting in surgery or limiting function for greater than 6 weeks
- 4) Injuries that would limit performance in this study
- 5) Diagnosed with a physical or psychological condition that would preclude functional testing (e.g. cardiac condition, clotting disorder, pulmonary condition)
- 6) Uncorrected visual or hearing impairment(s)
- 7) Require use of an assistive device
- 8) Unhealed wounds (cuts/abrasions) that would prevent CDO use
- 9) BMI > 35
- 10) Pregnancy

## Design and Methods:

Personal/demographic and anthropometric information will be used to fully characterize the study participants. We will collect multiple variables that have been previously associated with outcomes, including race, ethnicity, and education to characterize the cohort. Anthropometric and demographic information, such as age, biological sex, height, weight, leg length, shoe type, shoe length and width will also be used to characterize the cohort.

Patient-reported outcomes questionnaires will be used to evaluate participant pain and comfort and smoothness. Comfort and smoothness will be assessed using a modified version of the Socket Comfort Score, a reliable, valid, and sensitive measure of device fit and comfort.[3] These measures have been shown to effectively capture patient perception, are responsive to simple modifications to CDO device function, and will be applied in a manner consistent with a prior publication by the research team.[1] Participant will be asked to report their pain using a standard 11-point numerical pain rating scale, in which 0 = no pain and 10 = worst pain imaginable, at the start of session and at multiple points during testing.[4, 5] Semi-structured interviews will also be used to fully capture the participants perspectives, experience, and opinions associated with the study testing conditions.

Physical performance measures provide an objective and responsive assessment of an individual's functional mobility. Activities of daily life require performance of a range of functional tasks that require balance, agility, speed, and power. The four square step test (4SST) is a standardized and widely used test of functional mobility that requires rapid changes in direction that are often problematic following lower limb injury. The measure has good to excellent reliability and validity across multiple patient populations and groups and is a key dependent measure in most CDO-related studies to date and has demonstrated ability to detect changes in function in individuals with limb trauma and CDOs.[6-8, 9] The sit to stand 5 times (STS5) test is a well-established measure of lower limb muscle strength, endurance, and mobility.[10] The STS5 test has excellent reliability and good validity across a broad range of patient populations.[10-20]

Ground reaction force and motion capture data will be used to evaluate the motion and loading of the lower limb as participants walk on an over ground walkway at self-selected speed and a controlled speed based on leg length. [21, 22] The ability to collect reliable data across sites has been previously

demonstrated.[23] Previously established methods will be used to assess lower limb motion and moments.[22]

# **Statistical Analysis Plan**

## Analysis Methods:

All the primary dependent variables will be evaluated using similar statistical approaches within each group. One-way repeated measure ANOVAs will be used to evaluate the effect of CDO alignment. Paired t-tests with Bonferroni-Holm correction will be used for post-hoc comparisons. Multiple trials will be collected for each condition during testing.

# Power Analysis:

The number of participants proposed for this study are consistent with those from prior investigations by Dr. Wilken related to CDO design. Thirteen participants was sufficient to detect differences associated with AFO stiffness in a recent study by Dr. Wilken (PMID: 25193884).

## **Literature Cited:**

- 1. Ikeda, A.J., J.R. Fergason, and J.M. Wilken, Effects of altering heel wedge properties on gait with the Intrepid Dynamic Exoskeletal Orthosis. Prosthet Orthot Int, 2018. 42(3): p. 265-274
- 2. Rivera, J.C., et al., Posttraumatic osteoarthritis caused by battlefield injuries: the primary source of disability in warriors. J Am Acad Orthop Surg, 2012. 20 Suppl 1: p. S64-9.
- 3. Hanspal, R.S., K. Fisher, and R. Nieveen, Prosthetic socket fit comfort score. Disabil Rehabil, 2003. 25(22): p. 1278-80.
- 4. Hjermstad, M.J., et al., Studies comparing Numerical Rating Scales, Verbal Rating Scales, and Visual Analogue Scales for assessment of pain intensity in adults: a systematic literature review. J Pain Symptom Manage, 2011. 41(6): p. 1073-93.
- 5. Williamson, A. and B. Hoggart, Pain: a review of three commonly used pain rating scales. J Clin Nurs, 2005. 14(7): p. 798-804.
- 6. Patzkowski, J.C., et al., Comparative effect of orthosis design on functional performance. J Bone Joint Surg Am, 2012. 94(6): p. 507-15.
- 7. Bedigrew, K.M., et al., Can an integrated orthotic and rehabilitation program decrease pain and improve function after lower extremity trauma? Clin Orthop Relat Res, 2014. 472(10): p. 3017-25.
- 8. Hsu, J.R., et al., Patient Response to an Integrated Orthotic and Rehabilitation Initiative for Traumatic Injuries: The PRIORITI-MTF Study. J Orthop Trauma, 2017. 31 Suppl 1: p. S56-S62.
- 9. Dite, W. and V.A. Temple, A clinical test of stepping and change of direction to identify multiple falling older adults. Arch Phys Med Rehabil, 2002. 83(11): p. 1566-71.
- 10. Whitney, S.L., et al., Clinical measurement of sit-to-stand performance in people with balance disorders: validity of data for the Five-Times-Sit-to-Stand Test. Phys Ther, 2005. 85(10): p. 1034-45.
- 11. Beninato, M., L.G. Portney, and P.E. Sullivan, Using the International Classification of Functioning, Disability and Health as a framework to examine the association between falls and clinical assessment tools in people with stroke. Phys Ther, 2009. 89(8): p. 816-25.
- 12. Bohannon, R.W., Reference values for the five-repetition sit-to-stand test: a descriptive meta-analysis of data from elders. Percept Mot Skills, 2006. 103(1): p. 215-22.
- 13. Duncan, R.P., A.L. Leddy, and G.M. Earhart, Five times sit-to-stand test performance in Parkinson's disease. Arch Phys Med Rehabil, 2011. 92(9): p. 1431-6.
- 14. Lin, Y.C., R.C. Davey, and T. Cochrane, Tests for physical function of the elderly with knee and hip osteoarthritis. Scand J Med Sci Sports, 2001. 11(5): p. 280-6.
- 15. Mong, Y., T.W. Teo, and S.S. Ng, 5-repetition sit-to-stand test in subjects with chronic stroke: reliability and validity. Arch Phys Med Rehabil, 2010. 91(3): p. 407-13.
- 16. Newcomer, K.L., H.E. Krug, and M.L. Mahowald, Validity and reliability of the timed-stands test for patients with rheumatoid arthritis and other chronic diseases. J Rheumatol, 1993. 20(1): p. 21-7.
- 17. Paul, S.S., et al., Reproducibility of measures of leg muscle power, leg muscle strength, postural sway and mobility in people with Parkinson's disease. Gait Posture, 2012. 36(3): p. 639-42.
- 18. Schaubert, K.L. and R.W. Bohannon, Reliability and validity of three strength measures obtained from community-dwelling elderly persons. J Strength Cond Res, 2005. 19(3): p. 717-20.
- 19. Wang, T.H., H.F. Liao, and Y.C. Peng, Reliability and validity of the five-repetition sit-to-stand test for children with cerebral palsy. Clin Rehabil, 2012. 26(7): p. 664-71.

- 20. Wilken, J.M., et al., Physical performance assessment in military service members. J Am Acad Orthop Surg, 2012. 20 Suppl 1: p. S42-7.
- 21. Vaughan, C.L. and M.J. O'Malley, Froude and the contribution of naval architecture to our understanding of bipedal locomotion. Gait Posture, 2005. 21(3): p. 350-62.
- 22. Wilken, J.M., et al., Reliability and Minimal Detectible Change values for gait kinematics and kinetics in healthy adults. Gait Posture, 2012. 35(2): p. 301-7.
- 23. Kaufman, K., et al., Reliability of 3D gait data across multiple laboratories. Gait Posture, 2016. 49: p. 375-381.